CLINICAL TRIAL: NCT02102646
Title: MRI Substudy; Metabolic Changes Due to Iatrogenic Hypogonadism in Patients With Prostate Cancer: Orchiectomy vs. Triptorelin
Brief Title: MRI Substudy; Metabolic Changes Due to Iatrogenic Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Peter Busch Østergren, MD, Herlev Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kk2013 MRI
Record Dates: First submitted 2014-03-27; First posted 2014-04-03 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer; Metabolic Syndrome; Hypogonadism; Fatty Liver
MeSH Terms: conditions — Prostatic Neoplasms; Metabolic Syndrome; Hypogonadism; Fatty Liver | interventions — Triptorelin Pamoate; Orchiectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triptorelin (Active Comparator): Triptorelin 22,5mg/24th week intramuscularly
  Interventions: Drug: Triptorelin
- orchiectomy (Active Comparator): Androgen deprivation therapy by bilateral subcapsular orchiectomy
  Interventions: Procedure: Orchiectomy

INTERVENTIONS:
Drug: Triptorelin — Androgen deprivation therapy by Pamorelin 22,5mg/24 weeks administered intramuscularly.
  Other Names: Pamorelin
  Arms: Triptorelin
Procedure: Orchiectomy — Androgen deprivation therapy by bilateral subcapsular orchiectomy
  Other Names: Subcapsular orchiectomy
  Arms: orchiectomy

SUMMARY:
The purpose of this study is to investigate if androgen deprivation therapy in men with prostate cancer increases hepatic fat content and changes visceral/subcutaneous fat distribution.

DETAILED DESCRIPTION:
This is a substudy of the ongoing randomized trial entitled: Metabolic Changes Due to Iatrogenic Hypogonadism in Patients With Prostate Cancer: Orchiectomy vs. Triptorelin (EudraCT number: 2013-002553-29). 20 consecutive patients are anticipated to participate regardless of assignment to either orchiectomy or triptorelin.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for inclusion are patients who are included in the already ongoing Randomised trial entitled: Metabolic Changes Due to Iatrogenic Hypogonadism in Patients With Prostate Cancer: Orchiectomy vs. Triptorelin (EudraCT number: 2013-002553-29)

Exclusion Criteria:

* Implanted devices or foreign metallic bodies incompatible with Magnetic Resonance Imaging.
* claustrophobia
* Severe Psychiatric disease

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in hepatic fat content | At baseline (within 4 weeks of commencement of androgen deprivation therapy) and after 24 weeks
  Change in hepatic fat content measured by Magnetic Resonance Spectroscopy

SECONDARY OUTCOMES:
Change in visceral/subcutaneous fat mass | At baseline (within 4 weeks of commencement of androgen deprivation therapy) and after 24 weeks
  Changes in visceral and subcutaneous fat mass measured by Magnetic Resonance Imaging.
Correlation between Hepatic fat content and baseline androgen status | Androgen status measured before commencement of androgen deprivation therapy (ADT), hepatic fat content measured at baseline (within 1 month of commencing androgen deprivation therapy)
  To investigate possible correlation between androgen status before commencing androgen deprivation therapy and hepatic fat content at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Østergren, MD, Principal Investigator — Department of Urology, Herlev Hospital, Denmark
Locations (1):
- Herlev Hospital, Herlev, Denmark